CLINICAL TRIAL: NCT03135275
Title: MULTivessel Immediate Versus STAged RevaScularization in Acute Myocardial Infarction - The MULTISTARS AMI Trial
Brief Title: MULTivessel Immediate Versus STAged RevaScularization in Acute Myocardial Infarction -The MULTISTARS AMI Trial
Acronym: MULTISTARS AMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MULTISTARS_USZ
Record Dates: First submitted 2017-04-10; First posted 2017-05-01 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: ST-elevation Myocardial Infarction; Multivessel Coronary Disease
Keywords: ST-elevation Myocardial Infarction; Multivessel coronary disease; Immediate complete coronary revascularization; Staged complete coronary revascularization; Percutaneous coronary intervention; Biodegradable-polymer everolimus-eluting stent
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Staged complete PCI (Active Comparator): Patients randomized to staged complete PCI will have treated during the index admission only the culprit lesion and they will be hospitalized after 19-45 days, to complete the coronary revascularization on all the other significant coronary lesions. All the revascularizations will be performed with Synergy™ stent.
  Interventions: Procedure: Staged complete PCI; Device: Synergy™ stent
- Immediate complete PCI (Experimental): Patients randomized to immediate complete PCI will have treated immediately after the revascularization of the culprit lesion during the index procedure all the other significant coronary lesions. All the revascularizations will be performed with Synergy™ stent.
  Interventions: Procedure: Immediate complete PCI; Device: Synergy™ stent

INTERVENTIONS:
Procedure: Staged complete PCI — During the index procedure, patients will have treated with primary PCI the culprit lesion only. Patients will be hospitalized again after 19-45 days to undergo PCI of all the other significant coronary lesions. All the revascularizations will be performed with Synergy™ stent.
  Arms: Staged complete PCI
Procedure: Immediate complete PCI — During the index procedure, patients will have treated with primary PCI the culprit lesion, as well as all the other significant coronary lesions. All the revascularizations will be performed with Synergy™ stent.
  Arms: Immediate complete PCI
Device: Synergy™ stent — Bioabsorbable Polymer Drug-Eluting Stent

SUMMARY:
The primary objective of the trial is to compare, in patients presenting with ST segment elevation myocardial infarction (STEMI) and multi-vessel disease (MVD), the safety and efficacy of immediate complete revascularization of all significant coronary lesions versus culprit vessel only revascularization and staged percutaneous coronary intervention (PCI) of all significant coronary lesions (within 19 to 45 days), in a non-inferiority trial using a third generation, biodegradable-polymer, everolimus-eluting stent.

DETAILED DESCRIPTION:
An investigator-initiated, randomized, multicenter, two-arm, open-label study of consecutive patients presenting with STEMI and MVD in stable hemodynamic conditions, undergoing after successful PCI of the culprit lesion either (1:1 randomization) immediate revascularization of all additional target lesions during the index procedure or staged PCI of all additional target lesions (within 19 to 45 days) using the Boston Scientific Synergy™ stent.

The goal of this trial is to compare two treatment strategies that are currently performed in clinical practice: immediate complete revascularization versus staged complete revascularization in patients with STEMI and MVD.

Patients randomized to immediate complete revascularization will have treated during the index procedure, after revascularization of the culprit lesion, all significant non-culprit coronary lesions.

Patients randomized to staged complete revascularization will have treated during the index procedure only the culprit lesion, and they will be hospitalized after 19-45 days for complete revascularization of all significant non-culprit coronary lesions.

For both groups, lesion are considered significant when causing a ≥70% diameter stenosis by visual estimation in at least two projections on the coronary angiogram.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Spontaneous acute STEMI (patients presenting within 24 hours of symptom onset)
* Suitability for PCI from femoral or radial access
* Coronary anatomy suitable for complete coronary revascularization with Synergy® stent implantation
* Identifiable culprit lesion/artery
* At least one non-culprit coronary stenosis ≥ 70% in at least two projections, in a vessel with a lumen diameter ≥2.25 - ≤5.75 mm, other than the culprit artery
* TIMI Flow 3 or TIMI flow 2 after revascularization of the culprit artery
* Stable hemodynamics at the end of the culprit vessel revascularization

Exclusion Criteria:

* Inability to give informed consent
* Cardiogenic shock
* Prolonged resuscitation >10 min
* General unsuitability for PCI
* Need for emergency CABG
* Previous CABG
* Planned hybrid revascularization
* Coronary artery dissection
* STEMI due to ST
* Previous documented allergic reaction to everolimus or to any stent material
* Severe mechanical complication of acute myocardial infarction
* Pre-existing severe renal failure (eGFR <30 mL/min) or renal replacement therapy
* Chronic total occlusion of a major coronary artery
* Left main stem stenosis ≥50% or left main stem equivalent (ostial left anterior descending and ostial circumflex stenosis ≥70%)
* In-stent restenosis
* Panned coronary, cerebrovascular, or peripheral arterial revascularization
* Planned cardiac or major surgery
* Any contraindications for dual antiplatelet therapy with aspirin and a P2Y12 Inhibitor for at least 90 days, except for patients on oral anticoagulation
* Known pregnancy at the time of inclusion
* Participation in another clinical study with an investigational product
* Life expectancy <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2023-05 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is a composite of all-cause death, non-fatal myocardial infarction, unplanned ischemia-driven revascularization, hospitalization for heart failure, and stroke at 1 year | 1-year

SECONDARY OUTCOMES:
All-cause death, non-fatal myocardial infarction, unplanned ischemia-driven revascularization, hospitalization for heart failure, and stroke | 6 months
  Primary endpoint
All-cause death | 6 months, 1 year
  Single components of the primary endpoint
Non-fatal myocardial infarction | 6 months, 1 year
  Single components of the primary endpoint
Unplanned ischemia-driven revascularization | 6 months, 1 year
  Single components of the primary endpoint
Hospitalization for heart failure | 6 months, 1 year
  Single components of the primary endpoint
Stroke | 6 months, 1 year
  Single components of the primary endpoint
Target lesion revascularization (TLR) | 6 months, 1 year
Target vessel revascularization (TVR) | 6 months, 1 year
Non-cardiovascular death | 6 months, 1 year
Cardiac death | 6 months, 1 year
Cardiovascular death | 6 months, 1 year
Cardiac death or myocardial infarction | 6 months, 1 year
All-cause death or myocardial infarction | 6 months, 1 year
Stent thrombosis | 6 months, 1 year
Acute renal insufficiency or dialysis | 6 months, 1 year
Procedural success | 6 months, 1 year
Bleeding event (BARC definition) | 6 months, 1 year
Quality of life (EQ-5D questionnaire) | 6 months, 1 year

OTHER OUTCOMES:
Cost-effectiveness analysis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Barbara E. Stähli, MD, eMBA, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zürich, Cardiology Department, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wald DS, Morris JK, Wald NJ, Chase AJ, Edwards RJ, Hughes LO, Berry C, Oldroyd KG; PRAMI Investigators. Randomized trial of preventive angioplasty in myocardial infarction. N Engl J Med. 2013 Sep 19;369(12):1115-23. doi: 10.1056/NEJMoa1305520. Epub 2013 Sep 1. PMID 23991625
- [Background] Gershlick AH, Khan JN, Kelly DJ, Greenwood JP, Sasikaran T, Curzen N, Blackman DJ, Dalby M, Fairbrother KL, Banya W, Wang D, Flather M, Hetherington SL, Kelion AD, Talwar S, Gunning M, Hall R, Swanton H, McCann GP. Randomized trial of complete versus lesion-only revascularization in patients undergoing primary percutaneous coronary intervention for STEMI and multivessel disease: the CvLPRIT trial. J Am Coll Cardiol. 2015 Mar 17;65(10):963-72. doi: 10.1016/j.jacc.2014.12.038. PMID 25766941
- [Background] Engstrom T, Kelbaek H, Helqvist S, Hofsten DE, Klovgaard L, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, Clemmensen P, De Backer O, Ravkilde J, Tilsted HH, Villadsen AB, Aaroe J, Jensen SE, Raungaard B, Kober L; DANAMI-3-PRIMULTI Investigators. Complete revascularisation versus treatment of the culprit lesion only in patients with ST-segment elevation myocardial infarction and multivessel disease (DANAMI-3-PRIMULTI): an open-label, randomised controlled trial. Lancet. 2015 Aug 15;386(9994):665-71. doi: 10.1016/s0140-6736(15)60648-1. PMID 26347918
- [Background] Kornowski R, Mehran R, Dangas G, Nikolsky E, Assali A, Claessen BE, Gersh BJ, Wong SC, Witzenbichler B, Guagliumi G, Dudek D, Fahy M, Lansky AJ, Stone GW; HORIZONS-AMI Trial Investigators. Prognostic impact of staged versus "one-time" multivessel percutaneous intervention in acute myocardial infarction: analysis from the HORIZONS-AMI (harmonizing outcomes with revascularization and stents in acute myocardial infarction) trial. J Am Coll Cardiol. 2011 Aug 9;58(7):704-11. doi: 10.1016/j.jacc.2011.02.071. PMID 21816305
- [Background] Cavender MA, Milford-Beland S, Roe MT, Peterson ED, Weintraub WS, Rao SV. Prevalence, predictors, and in-hospital outcomes of non-infarct artery intervention during primary percutaneous coronary intervention for ST-segment elevation myocardial infarction (from the National Cardiovascular Data Registry). Am J Cardiol. 2009 Aug 15;104(4):507-13. doi: 10.1016/j.amjcard.2009.04.016. Epub 2009 Jun 18. PMID 19660603
- [Background] Widimsky P, Holmes DR Jr. How to treat patients with ST-elevation acute myocardial infarction and multi-vessel disease? Eur Heart J. 2011 Feb;32(4):396-403. doi: 10.1093/eurheartj/ehq410. Epub 2010 Nov 30. PMID 21118854
- [Background] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] Sabate M, Raber L, Heg D, Brugaletta S, Kelbaek H, Cequier A, Ostojic M, Iniguez A, Tuller D, Serra A, Baumbach A, von Birgelen C, Hernandez-Antolin R, Roffi M, Mainar V, Valgimigli M, Serruys PW, Juni P, Windecker S. Comparison of newer-generation drug-eluting with bare-metal stents in patients with acute ST-segment elevation myocardial infarction: a pooled analysis of the EXAMINATION (clinical Evaluation of the Xience-V stent in Acute Myocardial INfArcTION) and COMFORTABLE-AMI (Comparison of Biolimus Eluted From an Erodible Stent Coating With Bare Metal Stents in Acute ST-Elevation Myocardial Infarction) trials. JACC Cardiovasc Interv. 2014 Jan;7(1):55-63. doi: 10.1016/j.jcin.2013.07.012. Epub 2013 Dec 11. PMID 24332419
- [Result] Stahli BE, Varbella F, Linke A, Schwarz B, Felix SB, Seiffert M, Kesterke R, Nordbeck P, Witzenbichler B, Lang IM, Kessler M, Valina C, Dibra A, Rohla M, Moccetti M, Vercellino M, Gaede L, Bott-Flugel L, Jakob P, Stehli J, Candreva A, Templin C, Schindler M, Wischnewsky M, Zanda G, Quadri G, Mangner N, Toma A, Magnani G, Clemmensen P, Luscher TF, Munzel T, Schulze PC, Laugwitz KL, Rottbauer W, Huber K, Neumann FJ, Schneider S, Weidinger F, Achenbach S, Richardt G, Kastrati A, Ford I, Maier W, Ruschitzka F; MULTISTARS AMI Investigators. Timing of Complete Revascularization with Multivessel PCI for Myocardial Infarction. N Engl J Med. 2023 Oct 12;389(15):1368-1379. doi: 10.1056/NEJMoa2307823. Epub 2023 Aug 27. PMID 37634190
- [Derived] Jakob P, Varbella F, Linke A, Schwarz B, Felix SB, Seiffert M, Kesterke R, Nordbeck P, Witzenbichler B, Lang IM, Kessler M, Valina C, Dibra A, Rohla M, Moccetti M, Vercellino M, Gaede L, Bott-Flugel L, Stehli J, Candreva A, Paneni F, Templin C, Schindler M, Wischnewsky M, Zanda G, Quadri G, Mangner N, Toma A, Magnani G, Clemmensen P, Luscher TF, Munzel T, Schulze PC, Laugwitz KL, Rottbauer W, Huber K, Neumann FJ, Schneider S, Riemer T, Weidinger F, Achenbach S, Richardt G, Kastrati A, Ford I, Ruschitzka F, Stahli BE; MULTISTARS A. M. I. Investigators. Impact of diabetes on outcomes of patients with ST-segment elevation myocardial infarction and multivessel coronary artery disease undergoing percutaneous coronary intervention. Clin Res Cardiol. 2025 Sep 10. doi: 10.1007/s00392-025-02745-x. Online ahead of print. PMID 40928512
- See also: Press release University Hospital Zurich — https://www.usz.ch/medienmitteilung-herzkranzgefaesse-sofort-erweitern/